CLINICAL TRIAL: NCT04196114
Title: Study on Feasibility of Targeted Epidural Spinal Stimulation to Improve MObility Recovery in Patients With Sub-acute Spinal Cord Injury
Brief Title: Study on Feasibility of Stimulation on the Lumbar Part of the Spinal Cord to Improve Mobility Recovery in Patients With Sub-acute Spinal Cord Injury
Acronym: STIMO-2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on-hold before first recruitment
Sponsor: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Principal Investigator, Jocelyne Bloch, Coordinating investigator, Ecole Polytechnique Fédérale de Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STIMO-2
Record Dates: First submitted 2019-12-05; First posted 2019-12-12 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All patients implanted.
  Interventions: Device: STIMO-2 device implantation

INTERVENTIONS:
Device: STIMO-2 device implantation — Implantation of SCS lead in epidural space and implantation of neurostimulator in abdominal region

SUMMARY:
The STIMO-2 study aims to investigate TESS-supported rehabilitation training in sub-acute spinal cord injury (< 6 months post-injury). The primary endpoint of this study is to assess the safety and feasibility of TESS. The preliminary effectiveness of the therapy is the secondary study endpoint. The mobility recovery status of patients, who undergo TESS-supported rehabilitation, will be assessed at 12 months post SCI, compared to their predicted recovery expectations based on standard rehabilitation program

ELIGIBILITY:
Inclusion criteria (non-exhaustive list)

* Patient enrolled in the EMSCI study
* Age 18 to 70 years old included
* Focal spinal cord injury due to trauma
* Patient with history of SCI within the past 6 months (sub-acute SCI)
* Vertebral lesion T11 or above
* Psychological condition compatible with study participation
* Able and willing to fulfil all study procedures

Exclusion criteria (non-exhaustive list)

* Severe or chronic medical disorder pre-existing SCI affecting rehabilitation
* Active implanted device such as a pacemaker, implantable cardiac defibrillator
* Inability to follow study procedures, e.g. due to language problems, psychological disorders, dementia
* Pregnant or breast feeding
* Participation in other interventional study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety Measure: occurence of Serious Adverse Event | Through study completion, until 12 months after injury
  Occurrence of Serious Adverse Event that are deemed related or possibly related to study procedure or to study investigational system
Feasibility Measure: use of TESS stimulation (in minutes) for improved mobility | Through study completion, until 12 months after injury
  Measure of the absolute and relative usage of TESS (in minutes) during mobility rehabilitation sessions.

SECONDARY OUTCOMES:
Preliminary effectiveness: assessment of function recovery of leg motor function using the 6 mnWT distance | Through study completion, until 12 months after injury
  This endpoint will compare each patient's 6mnWT distance at 12 months post Date Of Injury to historical controls.
Preliminary effectiveness: mobility assessment using SCIM-III mobility score | Through study completion, until 12 months after injury
  This endpoint will compare each patient's SCIM-III mobility score at 12 months post Date Of Injury to historical controls.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No